CLINICAL TRIAL: NCT05653596
Title: Virtual Reality-Based Cognitive Intervention for Women With Cognitive Complaints Following Breast Cancer Treatment
Brief Title: VR-based Intervention for Cognitive Restoration
Acronym: CHEERS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chungnam National University (Other)
Responsible Party: Principal Investigator, Mi Sook Jung, Associate professor, Chungnam National University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ChungnamNU.J1
Record Dates: First submitted 2022-12-07; First posted 2022-12-16 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Cognitive Dysfunction; Virtual Reality
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: VR restorative intervention (Experimental): Individuals who are assigned to the experimental group will receive a 4-week VR-based cognitive intervention.
  Interventions: Behavioral: Virtual reality-based cognitive intervention
- Control: Usual care (No Intervention): Individuals who are assigned to the control group will receive the usual care and then receive the same intervention as they wish.

INTERVENTIONS:
Behavioral: Virtual reality-based cognitive intervention — This intervention consists of 12 different VR contents that were developed for this trial. Each content includes 10-12 scenes with visual and auditory stimuli generated from nature. Participants will view 3D nature videos using a VR headset for 20 minutes every other day, three times per week for one month.
  Arms: Experimental: VR restorative intervention

SUMMARY:
The aim of this study is to test the efficacy of a nature-based cognitive intervention to restore cognitive function among women treated for breast cancer.

DETAILED DESCRIPTION:
Cognitive dysfunction is a kind of cluster of commonly reported neurotoxic symptoms following cancer diagnosis and treatment, especially chemotherapy. Our previous studies found that breast cancer patients and survivors had greater difficulties in performing attention, working memory, and executive function tasks and had persistent neural inefficiency of an executive network of the brain than disease and treatment counterparts.

The aim of this study is to test the efficacy of a nature-based cognitive intervention to restore cognitive function among women with cognitive complaints after breast cancer treatment. All participants will receive the initial screening to verify their cognitive status and then will be randomly assigned to the experimental or control group. The experimental group will receive a 4-week cognitive intervention by using a VR headset. Each VR content includes 10-12 video scenes with visual and auditory stimuli that were generated from nature.

ELIGIBILITY:
Inclusion Criteria:

* Being treated with chemotherapy for breast cancer
* Having affirmative responses to three questions about cognitive problems and their impact on daily performance
* Having FACT-Cog scores of 58 or less
* Having Mini-Cog scores of 3 and higher
* Having the ability to read, understand or respond to questionnaires and cognitive assessment
* Being willing to participate and able to provide written informed consent

Exclusion Criteria:

* Having metastatic breast cancer
* Having Patient Health Questionnaire-2 score of 3 and higher
* Being diagnosed with neurological disorders such as dementia, multiple sclerosis, or traumatic brain injury
* Having epilepsy or seizure
* Having 'quite a bit' or 'extremely' severe level of nausea and vomiting
* Having visual or hearing impairments
* Having other problems that prevent them from wearing the VR headset

Ages: 19 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Central Nervous System Vital Signs (CNSVS) | Cognitive function will be assessed at baseline
  The CNSVS will be used to assess global and domain-specific cognitive function
Central Nervous System Vital Signs (CNSVS) | Cognitive function will be assessed at 4 weeks after baseline (immediate post-intervention)
  The CNSVS will be used to assess global and domain-specific cognitive function
Central Nervous System Vital Signs (CNSVS) | Cognitive function will be assessed at 8 weeks after baseline (4 weeks after intervention)
  The CNSVS will be used to assess global and domain-specific cognitive function
Functional Assessment of Cancer Therapy-Cognitive | Perceived cognitive function will be assessed at baseline
  The FACT-Cog will be used to assess self-reported effectiveness in cognitive function
Functional Assessment of Cancer Therapy-Cognitive | Perceived cognitive function will be assessed at 4 weeks after baseline (immediate post-intervention)
  The FACT-Cog will be used to assess self-reported effectiveness in cognitive function
Functional Assessment of Cancer Therapy-Cognitive | Perceived cognitive function will be assessed at 8 weeks after baseline (4 weeks after intervention)
  The FACT-Cog will be used to assess self-reported effectiveness in cognitive function

SECONDARY OUTCOMES:
Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) | Fatigue will will be assessed at baseline, 4 weeks (immediate post-intervention), and 8 weeks (4 weeks after intervention)
  The FACIT-F will be used to assess experience and impact of fatigue
Patient Health Questionnaire (PHQ) | Depression will be assessed at baseline, 4 weeks (immediate post-intervention), and 8 weeks (4 weeks after intervention)
  The PHQ will be used to assess depressed mood
Pittsburgh Sleep Quality Index (PSQI) | Sleep problems will be assessed at baseline, 4 weeks (immediate post-intervention), and 8 weeks (4 weeks after intervention)
  The PSQI will be used to assess sleep problems
Functional Assessment of Cancer Therapy-General (FACT-G) | Quality of life will be assessed at baseline, 4 weeks (immediate post-intervention), and 8 weeks (4 weeks after intervention)
  The FACT-G will be used to assess health-related quality of life
Perceived Restorativeness for Activities Scale (PRAS) | Perceived restorativeness will be assessed at baseline, 4 weeks (immediate post-intervention), and 8 weeks (4 weeks after intervention)
  The PRAS will be used to assess perceived restorativeness of their activities engaged to improve cognition

CONTACTS AND LOCATIONS:
Overall Officials: Mi Sook Jung, PhD, Principal Investigator — Chungnam National University
Locations (1):
- Cognitive Health Education and Research Center, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No